CLINICAL TRIAL: NCT05965141
Title: A Phase II Prospective Single-arm Clinical Study of Aribulin Combined With Carboplatin and Bevacizumab in the First-line Treatment of Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: Aribulin Combined With Carboplatin and Bevacizumab in the Treatment of Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-LCYJ-YY01
Record Dates: First submitted 2023-04-23; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aribulin in combination with carboplatin and bevacizumab (Experimental): This is a one-arm study without randomization. There was only one trial group of Aribulin combined with carboplatin and bevacizumab.
  Interventions: Drug: Aribulin;carboplatin;bevacizumab

INTERVENTIONS:
Drug: Aribulin;carboplatin;bevacizumab — Aribulin combined with carboplatin and bevacizumab in first-line treatment of platinum-sensitive recurrent ovarian cancer.

SUMMARY:
This is a prospective phase II, single-center, single-arm clinical study of platinum-sensitive relapsed ovarian cancer. The main objective of this study is to evaluate the efficacy, safety and tolerability of Aribrine combined with carboplatin and bevacizumab in first-line treatment of platinum-sensitive relapsed ovarian cancer.

DETAILED DESCRIPTION:
This is a phase II prospective, single-center, single-arm clinical study for platinum-sensitive recurrent ovarian cancer. The main objective of this study is to evaluate the efficacy, safety and tolerability of alibulin combined with carboplatin and bevacizumab in first-line treatment of platinum-sensitive recurrent ovarian cancer.

Trial time plan: The inclusion time of the plan: 22 months. Planned trial duration: 24 months.

1. Experimental drugs: Aribrine mesylate injection, carboplatin, bevacizumab.
2. Administration regimen: Iribrine mesylate injection: 1.4mg/m2i.v. 30 min, d1 d8, every 21 days; Carboplatin: AUC=5~6 i.v. d1, every 21 days; Bevacizumab: 7.5mg/kg, i.v. 30-90 min,d1, every 21 days. The dose can be adjusted according to the state of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable or immeasurable disease (RECIST v1.1) or CA 125 evaluable disease (GCIG criteria) or histologically confirmed diagnosis of recurrent ovarian cancer.
* First disease recurrence after first-line platinum chemotherapy >6 months.
* 18 years of age ≤75 years of female.
* Expected survival ≥ 3 months.

Exclusion Criteria:

* Partial tumor related symptoms.
* Partial comorbidity.
* Subjects developed new secondary malignancies.
* other.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | During treatment, imaging examinations were performed ±3 days every 2 cycles and D0±1 days per cycle for CA-125. When the efficacy was evaluated as PR or CR, imaging was performed again at 6 weeks ±3 days.
  The proportion of subjects who achieved PR and CR.

SECONDARY OUTCOMES:
Disease control rate | During treatment, imaging examinations were performed ±3 days every 2 cycles and D0±1 days per cycle for CA-125. When the efficacy was evaluated as PR or CR, imaging was performed again at 6 weeks ±3 days.
  Percentage of subjects who achieved PR, CR, and SD.
Progression-free survival time | During treatment, imaging examinations were performed ±3 days every 2 cycles and D0±1 days per cycle for CA-125. When the efficacy was evaluated as PR or CR, imaging was performed again at 6 weeks ±3 days.
  The time between the patient's first treatment date and any recorded tumor progression or death from any cause.
Clinical benefit rate | During treatment, imaging examinations were performed ±3 days every 2 cycles and D0±1 days per cycle for CA-125. When the efficacy was evaluated as PR or CR, imaging was performed again at 6 weeks ±3 days.
  Percentage of subjects who achieved PR, CR, and SD for at least 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jingqi Chen, Study Chair — Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ren JS, Masuyer E, Ferlay J. Global estimates of cancer prevalence for 27 sites in the adult population in 2008. Int J Cancer. 2013 Mar 1;132(5):1133-45. doi: 10.1002/ijc.27711. Epub 2012 Jul 26. PMID 22752881
- [Background] Ramalingam P. Morphologic, Immunophenotypic, and Molecular Features of Epithelial Ovarian Cancer. Oncology (Williston Park). 2016 Feb;30(2):166-76. PMID 26892153
- [Background] Paik ES, Lee YY, Lee EJ, Choi CH, Kim TJ, Lee JW, Bae DS, Kim BG. Survival analysis of revised 2013 FIGO staging classification of epithelial ovarian cancer and comparison with previous FIGO staging classification. Obstet Gynecol Sci. 2015 Mar;58(2):124-34. doi: 10.5468/ogs.2015.58.2.124. Epub 2015 Mar 16. PMID 25798426
- [Background] Mahmood RD, Morgan RD, Edmondson RJ, Clamp AR, Jayson GC. First-Line Management of Advanced High-Grade Serous Ovarian Cancer. Curr Oncol Rep. 2020 Jun 4;22(6):64. doi: 10.1007/s11912-020-00933-8. PMID 32494876
- [Background] Coleman RL, Brady MF, Herzog TJ, Sabbatini P, Armstrong DK, Walker JL, Kim BG, Fujiwara K, Tewari KS, O'Malley DM, Davidson SA, Rubin SC, DiSilvestro P, Basen-Engquist K, Huang H, Chan JK, Spirtos NM, Ashfaq R, Mannel RS. Bevacizumab and paclitaxel-carboplatin chemotherapy and secondary cytoreduction in recurrent, platinum-sensitive ovarian cancer (NRG Oncology/Gynecologic Oncology Group study GOG-0213): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2017 Jun;18(6):779-791. doi: 10.1016/S1470-2045(17)30279-6. Epub 2017 Apr 21. PMID 28438473
- [Background] Jordan MA, Wilson L. Microtubules as a target for anticancer drugs. Nat Rev Cancer. 2004 Apr;4(4):253-65. doi: 10.1038/nrc1317. No abstract available. PMID 15057285
- [Background] Smith JA, Wilson L, Azarenko O, Zhu X, Lewis BM, Littlefield BA, Jordan MA. Eribulin binds at microtubule ends to a single site on tubulin to suppress dynamic instability. Biochemistry. 2010 Feb 16;49(6):1331-7. doi: 10.1021/bi901810u. PMID 20030375
- [Background] Ito K, Hamamichi S, Abe T, Akagi T, Shirota H, Kawano S, Asano M, Asano O, Yokoi A, Matsui J, Umeda IO, Fujii H. Antitumor effects of eribulin depend on modulation of the tumor microenvironment by vascular remodeling in mouse models. Cancer Sci. 2017 Nov;108(11):2273-2280. doi: 10.1111/cas.13392. Epub 2017 Sep 22. PMID 28869796
- [Background] Cortes J, Schoffski P, Littlefield BA. Multiple modes of action of eribulin mesylate: Emerging data and clinical implications. Cancer Treat Rev. 2018 Nov;70:190-198. doi: 10.1016/j.ctrv.2018.08.008. Epub 2018 Aug 21. PMID 30243063
- [Background] Hensley ML, Kravetz S, Jia X, Iasonos A, Tew W, Pereira L, Sabbatini P, Whalen C, Aghajanian CA, Zarwan C, Berlin S. Eribulin mesylate (halichondrin B analog E7389) in platinum-resistant and platinum-sensitive ovarian cancer: a 2-cohort, phase 2 study. Cancer. 2012 May 1;118(9):2403-10. doi: 10.1002/cncr.26569. Epub 2011 Sep 20. PMID 21935916
- [Background] Cortes J, O'Shaughnessy J, Loesch D, Blum JL, Vahdat LT, Petrakova K, Chollet P, Manikas A, Dieras V, Delozier T, Vladimirov V, Cardoso F, Koh H, Bougnoux P, Dutcus CE, Seegobin S, Mir D, Meneses N, Wanders J, Twelves C; EMBRACE (Eisai Metastatic Breast Cancer Study Assessing Physician's Choice Versus E7389) investigators. Eribulin monotherapy versus treatment of physician's choice in patients with metastatic breast cancer (EMBRACE): a phase 3 open-label randomised study. Lancet. 2011 Mar 12;377(9769):914-23. doi: 10.1016/S0140-6736(11)60070-6. Epub 2011 Mar 2. PMID 21376385
- [Background] Kaufman PA, Awada A, Twelves C, Yelle L, Perez EA, Velikova G, Olivo MS, He Y, Dutcus CE, Cortes J. Phase III open-label randomized study of eribulin mesylate versus capecitabine in patients with locally advanced or metastatic breast cancer previously treated with an anthracycline and a taxane. J Clin Oncol. 2015 Feb 20;33(6):594-601. doi: 10.1200/JCO.2013.52.4892. Epub 2015 Jan 20. PMID 25605862
- [Background] De Angelis C, Bruzzese D, Bernardo A, Baldini E, Leo L, Fabi A, Gamucci T, De Placido P, Poggio F, Russo S, Forestieri V, Lauria R, De Santo I, Michelotti A, Del Mastro L, De Laurentiis M, Giuliano M, De Placido S, Arpino G. Eribulin in combination with bevacizumab as second-line treatment for HER2-negative metastatic breast cancer progressing after first-line therapy with paclitaxel and bevacizumab: a multicenter, phase II, single arm trial (GIM11-BERGI). ESMO Open. 2021 Apr;6(2):100054. doi: 10.1016/j.esmoop.2021.100054. Epub 2021 Feb 16. PMID 33601296
- [Background] Hardy-Bessard AC, Brocard F, Clatot F, Lortholary A, You B, Grenier J, Martin-Babau J, Lucas B, Meunier J, Ferrero JM, Savoye AM, Marti A, Despax R, Moullet I, Emile G. First-line bevacizumab and eribulin combination therapy for HER2-negative metastatic breast cancer: Efficacy and safety in the GINECO phase II ESMERALDA study. Breast. 2020 Dec;54:256-263. doi: 10.1016/j.breast.2020.09.011. Epub 2020 Sep 30. PMID 33188992
- [Background] Yuan P, Hu X, Sun T, Li W, Zhang Q, Cui S, Cheng Y, Ouyang Q, Wang X, Chen Z, Hiraiwa M, Saito K, Funasaka S, Xu B. Eribulin mesilate versus vinorelbine in women with locally recurrent or metastatic breast cancer: A randomised clinical trial. Eur J Cancer. 2019 May;112:57-65. doi: 10.1016/j.ejca.2019.02.002. Epub 2019 Mar 29. PMID 30928806
- [Background] Zhao Y, Xie N, Li W, Chen W, Lv Z, Zheng Y, Sun T, Liu J, Zhang J, Hu S, Wang Y, Gong C, Li Y, Xie Y, Ge R, Xu F, Wang B. Real-world effectiveness of eribulin in heavily pretreated patients with metastatic breast cancer in China: a multicenter retrospective study. Ther Adv Med Oncol. 2021 Jul 9;13:17588359211030210. doi: 10.1177/17588359211030210. eCollection 2021. PMID 34290830